CLINICAL TRIAL: NCT02075268
Title: An Open Label, Single Dose Study to Characterize the Pharmacokinetics and Pharmacodynamics of Prasugrel in Healthy Male Adult Subjects
Brief Title: Clinical Trial to Characterize Pharmacokinetic-pharmacodynamic (PKPD) of Prasugrel 10 mg or 30 mg in Healthy Volunteers
Acronym: PRAS-AM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hyeong-Seok Lim, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PRAS-AM; 2014-0064 (Other: Institutional review board of Asan Medical Center)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Korean; Healthy; Male
MeSH Terms: interventions — Prasugrel Hydrochloride; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 10 mg, 30 mg (Other): To compare PKPD of prasugrel 10 or 30 mg, 4 subjects will be given 10 mg of prasugrel (one tablet of 10 mg of Effient) on day 1 as a single oral dose and another 4 subjects will be given 30 mg of prasugrel (3 tablets of 10 mg of Effient) on day 1 as a single oral dose.
  Interventions: Drug: prasugrel

INTERVENTIONS:
Drug: prasugrel — prausugrel 10 or 30 mg will be administrated as single dose under overnight fast.
  Other Names: Effient 10 mg tablet will be used as study drug.

SUMMARY:
An open label, parallel study to characterize the pharmacokinetics and pharmacodynamics of Prasugrel 30 mg or 60 mg in healthy male adult subjects

DETAILED DESCRIPTION:
1. Screening
2. Enrollment and treatment randomization
3. Confinement to Research Unit from day - 1 to day 2
4. Outpatient visit : 2 times ( 48 and 73 hours after dosing)
5. Drug administration : Overnight Fasting
6. Blood sampling for PK, PD and genotyping

   1. PK: up to 24 hours after dosing
   2. PD: up to 72 hours after dosing

ELIGIBILITY:
Inclusion Criteria:

* male aged 19 to 45 years
* weigh over 60 kg
* body mass index 18 to 30 kg/m2

Exclusion Criteria:

* any history or state of clinically significant disease
* any gastrointestinal disease may interfere absorption of drug
* any history of hypersensitivity to prasugrel or other drug
* any history of taking herbal medication within 30 days before dosing or taking prescription medication within 14 days before dosing or taking over the counter drug within 7 days before dosing
* taking investigational drug within 60 days before dosing
* transfused within 30 days or donated blood within 60 days before dosing
* Positive serology test ( Hepatitis B surface antigen (HBs Ag), HIV, HCV)
* Clinically significant finding in laboratory result or electrocardiogram result

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
plasma R-138727 and R-95913 concentrations | predose, 10 min, 15 min, 25 min, 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 4 h, 6 h, 8 h, 12 h and 24 h after dosing

SECONDARY OUTCOMES:
Maximal platelet aggregation | predose, 15 min, 0.5 h, 1 h, 2 h, 4 h, 8 h, 24 h, 48 h and 72 h after dosing
  Maximal platelet aggregation will be measured by light transmission test

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Jeon HS, Kim MJ, Choi HY, Kim YH, Kim EH, Kim AR, Park HJ, Bae KS, Lim HS. Pharmacokinetics and pharmacodynamics of ticagrelor and prasugrel in healthy male Korean volunteers. Clin Ther. 2015 Mar 1;37(3):563-73. doi: 10.1016/j.clinthera.2015.01.010. Epub 2015 Feb 16. PMID 25697420